CLINICAL TRIAL: NCT01134653
Title: Efficacy of Stretch Band Ankle Traction Technique in the Treatment of Acute Ankle Sprains.
Brief Title: A Comparison of Early Mobilization Versus Traditional Treatment for Acute Ankle Sprains.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Lindsay Alfano, Assistant Professor, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB07-00110; 663110 (Other Grant/Funding Number: Foundation for Physical Therapy)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Ankle Sprain
Keywords: Acute ankle sprain in children and young adults
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jump stretch (Experimental): Distraction with early mobilization
  Interventions: Other: Jump Stretch
- RICE (Active Comparator): Subject receive standard ankle sprain treatment of Rest Ice compression and elevation for one week. This is followed by traditional strength and range of motion therapy. The subject does not receive distraction treatments.
  Interventions: Other: Jump Stretch

INTERVENTIONS:
Other: Jump Stretch — distraction with early mobilization

SUMMARY:
Acute ankle sprain is one of the most common musculoskeletal injuries, accounting for an estimated 2 million injuries per year and 20% of all sports injuries in the United States. Ankle sprains can lead to prolonged periods of pain, difficulty with mobility, and lost work or play time. Current best practice guidelines for treatment of an acute ankle sprain are protection, rest, ice, compression and elevation (PRICE). However recent systematic reviews for ankle sprains call into question this treatment. Two critical components; immobilization and ice, have little or no evidence of efficacy for ankle sprain. Interestingly, mobilization appears to be more effective at reducing the pain, swelling and stiffness of musculoskeletal injuries including ankle sprains. Historically the limitation to early mobilization has been pain. Recently developed stretch bands have been introduced to the therapy market as a tool that allows pain-free active and resisted ankle movement after acute ankle sprain.

The investigators propose a double blind randomized controlled study to compare 2 ankle sprain treatments on their ability to speed recovery and reduce morbidities such as pain, swelling and weakness.

ELIGIBILITY:
Inclusion Criteria:

* 3 day post injury

Exclusion Criteria:

* fracture
* chronic sprain

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
days until return to activities | discharge
  days until return to activities

SECONDARY OUTCOMES:
VAS scale | 1 week
  scale to measure pain 1 week post enrollment
strength | 1 week
  change in strength
Figure of Eight Measurement | 1 week
  change in size of ankle in figure 8 measurement to swelling

CONTACTS AND LOCATIONS:
Overall Officials: Linda p Lowes, PhD, Principal Investigator — columbus cri
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States